CLINICAL TRIAL: NCT03316612
Title: The Effect of Vaccinium Myrtillus L. Extract Intake on Human Metabolism: A Randomized Double-Blind Trial
Brief Title: The Effect of Vaccinium Myrtillus L. Extract Intake on Human Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C01-201611090005
Record Dates: First submitted 2017-10-17; First posted 2017-10-20 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Healthy
Keywords: Advanced Glycation End Products, Metabolites, Gut Microbiota

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The all details of groups assignment are arranged and controlled by the research designers. The color, shape, and external packaging of the bilberry extract and placebo are consistent (brown oval tablets). Each bottle of tablets will be marked with the name (or identify number) of the participants by research designers. Thus, the grouping of participants is blind to the rest of the researchers (like outcomes assessors).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Ingredients: Vaccinium Myrtillus L. extracts, and excipients (cellulose microcrystalline, mannitol, silica, magnesium stearate, coating agent)
  Brown oval tablet, 650mg per tablet with 150mg Vaccinium Myrtillus L. extracts, twice a day, 2 tablets each time.
  The intervention period is about 3 months.
  Interventions: Dietary Supplement: Vaccinium Myrtillus L. extract
- Placebo group (Placebo Comparator): Ingredients: excipients (cellulose microcrystalline, mannitol, silica, magnesium stearate, coating agent)
  Brown oval tablet without Vaccinium Myrtillus L. extracts, 650mg per tablet, twice a day, 2 tablets each time.
  The intervention period is about 3 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vaccinium Myrtillus L. extract — Twice a day, 2 tablets each time. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Intervention group
Dietary Supplement: Placebo — Twice a day, 2 tablets each time. Do not take any other medicine, traditional Chinese medicine, or dietary supplements.
  Arms: Placebo group

SUMMARY:
Advanced glycation end-products (AGEs) has been linked to ageing, and many metabolic diseases. The findings of previous experiments suggested that the extracts from polyphenol-rich bilberry might inhibit the formation of AGEs. This is a randomized double-blind trial, aims to study the effect of Vaccinium Myrtillus L. natural extracts on AGEs and human metabolism. Firstly, we will investigate the efficacy of Bilberry extracts on lowering the levels of advanced glycation end-products (AGEs). Secondly, we will conduct 16S rRNA sequencing and ultra-high performance liquid chromatography-tandem mass spectrometric (UPLC-MS/MS) detection to explore the role of bilberry extracts on gut microbiota as well as metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years of age
* Able to give informed connect

Exclusion Criteria:

* Pregnancy
* Known cardiovascular disease (stroke, ischemic heart disease and so on), diabetes, hypertension and any other chronic disease.
* Known gastrointestinal disease, such as Irritable Bowel Syndrome(IBS), functional bowel disease and so on.
* Evidence of drug or alcohol abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma AGEs levels | At 0 week (baseline), 4th week, 10th week.
  Using UPLC-MS/MS to detect plasma AGEs (including CML, CEL, MG-H1).
Changes in urinary AGEs levels | At 0 week (baseline), 4th week, 10th week.
  Using UPLC-MS/MS to detect urinary AGEs (including CML, CEL, MG-H1).
Changes in plasma sRAGE levels | At 0 week (baseline), 4th week, 10th week.
  sRAGE (soluble Receptor for Advanced Glycation End-products)
Changes in transcription levels of RAGE and AGER1 | At 0 week (baseline), 4th week, 10th week.
  Extract and isolate peripheral blood mononuclear cells (PBMC) from participants. Using the PCR technology to detect the mRNA levels of RAGE and AGER1.
Changes in gut microbiota | At 0 week (baseline), 10th week.
Changes in plasma metabolites | At 0 week (baseline), 4th week, 10th week.

SECONDARY OUTCOMES:
Changes in skin AGEs levels | At 0 week (baseline), 4th week, 10th week.
  Using AGE Reader to quickly and noninbasively measure skin AGEs by means of fluorescence techniques.
Changes in body weight | At 0 week (baseline), 4th week, 10th week.
Change in body composition (body fat mass and lean mass) | At 0 week (baseline), 4th week, 10th week.
Changes in blood lipids profile | At 0 week (baseline), 4th week, 10th week.
  Fasting plasma Total cholesterol, Low Density Lipoprotein, High Density Lipoprotein and triglycerides.
Changes in pro-inflammatory markers | At 0 week (baseline), 4th week, 10th week.
  Fasting plasma C-reactive protein, interleukin-6 and tumor necrosis factor-α
Changes in fecal short chain fatty acids (SCFA) | At 0 week (baseline), 10th week.

CONTACTS AND LOCATIONS:
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided